CLINICAL TRIAL: NCT04058288
Title: Targeted Noninvasive Brain Stimulation (T-NIBS) for Improving Hand Dexterity in Stroke Patients
Brief Title: Targeted Noninvasive Brain Stimulation to Improve Hand Dexterity in Stroke Patients
Acronym: T-NIBS
Status: Completed | Type: Observational
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Vikram Shenoy Handiru, Associate Research Scientist, Kessler Foundation
Other Study IDs: R-1056-19
Record Dates: First submitted 2019-07-29; First posted 2019-08-15 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Stroke
Keywords: stroke; HD-tDCS; musicglove; Upper-limb rehab
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Stroke: People suffering from upper-limb motor dysfunction due to stroke
  Interventions: Device: High-definition Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: High-definition Transcranial Direct Current Stimulation — Stimulation sessions will be conducted on 2 different visits separated by 2-week gap. In a crossover design, Anodal HD-tDCS will be delivered either in Active/Sham mode (during the first visit) and Sham/Active during the second visit in a 4x1 ring configuration (center electrode being Anode and the surrounding 4 electrodes being cathodes) over the affected motor area.

SUMMARY:
This study will investigate the use of High-definition Transcranial Direct Current Stimulation (HD-tDCS) in the functional improvement of hand dexterity while performing music-assisted hand exercises.

DETAILED DESCRIPTION:
Stroke is a serious medical and health problem in the US, and most of the stroke patients suffer from upper-limb motor deficits including weakened hand dexterity. As upper-limb motor functions are crucial for most of the daily living activities, there is a need for effective intervention. The current therapeutic approaches involve intensive physical therapy training involving repetitive tasks which causes fatigue and lack of engagement in the patients. To address this issue, the investigators will investigate the combined use of individually targeted noninvasive brain stimulation (T-NIBS) using High-definition Transcranial Direct Current Stimulation (HD-tDCS) and music-assisted hand exercises using MusicGlove to modulate the neuroplasticity in the desired manner to observe functional changes in hand dexterity.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-75 years
* Clinically diagnosed with hemiparetic stroke (weakness on one side - either left or right side of the body)
* Have had a stroke for more than 6 months
* Have weakness in moving the fingers of the affected hand
* Able to understand and perform the instructions that are part of the tDCS-MusicGlove testing and intervention.
* Willing and able to participate in and travel to Kessler Foundation for the screening session, MRI session, and tDCS-MusicGlove sessions.
* Able to sit and be active for 1.5 hours during the session without cardiac, respiratory and/or pain disturbances as assessed during the screening visit.
* Able to provide informed consent.
* Medically stable and not planning for a major change in medications for at least 4 weeks

Exclusion Criteria:

* Unable to move the hand because of muscle stiffness (scoring 3 or more on the Ashworth scale)
* Have lost the sensation of hand movement
* Have a history of alcohol abuse and/or illicit drug use
* Have a history of smoking within the past 5 years
* Have a problem with the eyesight that would make it difficult to notice the changing instructions on a computer screen
* Currently enrolled in another research study that might affect this research study
* A history of epilepsy (including family members who are diagnosed with epilepsy)
* An active history of migraine or chronic headache
* A history of mental illness (e.g. schizophrenia, anxiety, depression, and PTSD)
* Past or current history of treated ringing in the ears known as tinnitus or severe hearing problems
* Have a tattoo with metal-based ink in the head or neck.
* Have severe skin damage on the scalp
* Afraid of confined spaces (claustrophobic)
* Have metallic implants, including intracranial electrodes, surgical clips, shrapnel or a pacemaker.
* Currently taking medications that increase the risk of seizures
* Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primarily, the stroke survivors from the New Jersey/New York City area. Although not restricted to any primary care clinic, we encourage participants from the Kessler Institute for Rehabilitation.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in the Nine-Hole Peg Test (NHPT) scores | baseline (at day 1), during testing visits (day 2 and day 3)- all within 2 weeks from the screening and consenting
  NHPT is a secondary outcome measure of finger dexterity that can be used in stroke patients with upper extremity motor deficits. It is considered to be a reliable measure of hand dexterity and recommended for inclusion in NIH toolbox Assessment of Neurological and Behavioral Function. NHPT requires participants to repeatedly place nine pegs into nine holes, one at a time, as quickly as possible and then remove them from the holes. The total time needed to complete the task is then recorded.
Changes in the Dexterity and Speed Test (DAST) scores | baseline (at day 1), during testing visits (day 2 and day 3)- all within 2 weeks from the screening and consenting
  DAST is exclusively developed for MusicGlove performance assessment and it is designed to evaluate how fast and accurately do the subjects respond to the sequence of music notes that continuously sped up.

SECONDARY OUTCOMES:
Changes in the Cortical Excitability using Motor Evoked Potentials (MEP) | baseline (at day 1), during testing visits (day 2 and day 3) - all within 2 weeks from the screening and consenting
  MEP outcome measures have become the norm in brain stimulation studies. We hypothesize that the MEP amplitude and latency before- and after-intervention would reveal more information about the neuroplasticity changes during motor recovery. The motor evoked potential (MEP) will be provided by twenty unconditioned stimuli (120% RMT).

CONTACTS AND LOCATIONS:
Overall Officials: Guang Yue, PhD, Study Director — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No